CLINICAL TRIAL: NCT01975207
Title: Comparison Study of Family Practice Interventions for Depression in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Addiction & Mental Health Strategic Clinical Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: AMH-SCN-01
Record Dates: First submitted 2013-10-29; First posted 2013-11-04 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (No Intervention): Patients will have information collected on their quality of life (QOL) at baseline (EuroQual 5-item measure - "EQ-5D"). Patients will be followed up at week 12 for a repeated measure of QOL and a score on the depression rating scale being used in this study (Patient Health Questionnaire-9 item version - "PHQ-9"). Individuals will also be asked on their health care access frequency (HCAF) at baseline and follow up.
- Group 2 (Experimental): Group #2. Screening for depression followed by treatment as usual: Patients will complete baseline measurements of their score on the PHQ-9, self-reported HCAF and QOL (EQ-5D) score.
  The PHQ-9 score will be given to the clinic staff who will then follow up with treatment as usual. Patients will be followed up at week 12 for self-reported HCAF,PHQ-9 and QOL scores.
  Interventions: Behavioral: Treatment as usual
- Group 3 (Experimental): Group #3 is Internet intervention: At baseline patients will complete QOL (EQ-5D), PHQ-9 scores, and self-reported HCAF. Those who score 10 or more on the PHQ-9 will be offered a guided internet-based intervention for the treatment of depression by the study staff. Patients will be followed up at week 12 for self-reported HCAF, PHQ-9 and QOL scores.
  Interventions: Behavioral: Internet Intervention
- Group 4 (Experimental): Depression Treatment Pathway: At baseline patients will complete PHQ-9, QOL (EQ-5D) scores, and self-reported HCAF. Those who score 10 or more on the PHQ-9 will be offered the specific treatment as determined by the Depression Pathway by the clinic physician. Whenever possible, this pathway will be integrated into the local clinic's electronic medical record system, for ease of administration by the clinic. Patients will be followed up at week 12 for self-reported HCAF, PHQ-9 and QOL (EQ-5D) scores.
  Interventions: Behavioral: Depression Treatment Pathway

INTERVENTIONS:
Behavioral: Treatment as usual — Participants will be treated as per clinic's standard treatment for depression.
  Arms: Group 2
Behavioral: Internet Intervention — One of the major treatments for mild-moderate depressive disorders is cognitive behavioural therapy (CBT). It has been possible to operationalize some of this treatment and internet-based approaches to this have been developed. The most widely examined was developed in Australia and is termed "MoodGYM" (https://moodgym.anu.edu.au/welcome). This program has been widely studied, and these studies have shown it is very effective for many individuals in family practice
  Other Names: Guided internet-based invtervention; Moodgym; On-line CBT
  Arms: Group 3
Behavioral: Depression Treatment Pathway — There has been a growing awareness in health care circles that certain high frequency, high cost addiction and mental health disorders may be best addressed via the systemic adoption of clinical pathways. A clinical pathway is defined as "a multidisciplinary outline of anticipated care, placed in an appropriate timeframe, to help a patient with a specific condition or set of symptoms move progressively through a clinical experience to positive outcomes." A clinical pathway incorporates guidelines, protocols and evidence informed best practice into everyday use for the patient and family.
  Arms: Group 4

SUMMARY:
To determine if treatment of significant depressive symptoms identified in individuals attending a family practice improves either psychiatric outcome, overall health care costs, or Quality of Life (QOL). Two previously developed treatment approaches - an internet-based approach and a comprehensive depression pathway - will be compared to two control groups (those who have treatment as usual after screening for depression and measurement of QOL, and a second control group who will have QOL data only collected). The investigators hope to help Alberta Health Services identify which approach is best as rapidly as possible so that the best approach can be implemented throughout the province of Alberta.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and above
* Cognitively capable of independently understanding and confirming their desire to take part

Exclusion Criteria:

* 18 and under
* Cognitively incapable of independently understanding and confirming their desire to take part

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1489 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05-05 (Actual); Study Completion 2015-05-05 (Actual)

PRIMARY OUTCOMES:
Reduction in depression scores in those patients who have one of the two treatment interventions | 12 weeks
  We expect a reduction in depression scores in those patients who have one of the two treatment interventions (Groups #3 and #4) over a 12-week period, compared to those who are screened for depression, but only receive treatment as usual (Group #2).

SECONDARY OUTCOMES:
Reduction in total health care costs | 12 weeks/12 months
  We expect a reduction in total health care costs in the two treatment groups compared both to those who are not screened for depression (Group #1) and those who are screened for depression, but only receive treatment as usual (Group #2). This will be a within-subject comparison for total health care costs in the 12-weeks prior to the index visit compared to the total health care costs in the 12-weeks following the index visit. Mid-term costs will also be compared between groups for the 12-month period following the index visit. Examples of costs included are the number of doctors visits, any ambulance rides or emergency room visits and lab tests. The data collected will not include any diagnosis or results and will only be used for economic analysis. This data will be owned by the University of Alberta, will not be saved in medical records and no one but the study staff will have access to the data unless authorized by a governement agency or ethics board.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H Silverstone, M.D., Principal Investigator — Alberta Health Services and University of Alberta; Katherine Rittenbach, PhD, Study Director — Alberta Health services

REFERENCES:
- [Background] Hickie IB, Davenport TA, Luscombe GM, Moore M, Griffiths KM, Christensen H. Practitioner-supported delivery of internet-based cognitive behaviour therapy: evaluation of the feasibility of conducting a cluster randomised trial. Med J Aust. 2010 Jun 7;192(S11):S31-5. doi: 10.5694/j.1326-5377.2010.tb03690.x. PMID 20528705
- [Derived] Yan C, Rittenbach K, Souri S, Silverstone PH. Cost-effectiveness analysis of a randomized study of depression treatment options in primary care suggests stepped-care treatment may have economic benefits. BMC Psychiatry. 2019 Aug 5;19(1):240. doi: 10.1186/s12888-019-2223-3. PMID 31382932